CLINICAL TRIAL: NCT04621253
Title: Interaction of Cytochrome P450 Inhibition With Metamizole Metabolism in Healthy Subjects
Brief Title: Inhibition Metamizole 2020
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-01404
Record Dates: First submitted 2020-10-26; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Drug-drug Interaction
Keywords: Metamizole; Inhibition; Cytochrome P450
MeSH Terms: conditions — Inhibition, Psychological | interventions — Dipyrone

STUDY DESIGN:
Intervention Model Description: Randomized cross-over treatment with 3 different sequences
Who Masked: Investigator
Masking Description: Ciprofloxacin, Fluconazole and Placebo Capsules were produced under good manufacturing practice conditions and randomized by the responsible pharmacist. The investigator received emergency envelops in case of severe adverse reactions connected to the pretreatment to unblind the study, however the pharmacist retained the detailed randomization plan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ciprofloxacin (Active Comparator): Day 1: 750 mg ciprofloxacin capsule in the morning and evening Day 2: 750 mg ciprofloxacin capsule in the morning and evening Day 3: 750 mg ciprofloxacin capsule in the morning and evening Day 4: Study day, 750 mg ciprofloxacin 1h prior to 1000 mg metamizole.
  Interventions: Drug: Novalgin
- Fluconazole (Active Comparator): Day 1: 400 mg fluconazole in the morning, placebo capsule in the evening Day 2: 200 mg fluconazole in the morning, placebo capsule in the evening Day 3: 200 mg fluconazole in the morning, placebo capsule in the evening Day 4: Study day, 200 mg fluconazole 1h prior to 1000 mg metamizole.
  Interventions: Drug: Novalgin
- Placebo (Placebo Comparator): Day 1: placebo capsule in the morning and evening Day 2: placebo capsule in the morning and evening Day 3: placebo capsule in the morning and evening Day 4: Study day, placebo capsule 1h prior to 1000 mg metamizole.
  Interventions: Drug: Novalgin

INTERVENTIONS:
Drug: Novalgin — Single dose of 1000 mg metamizole, 1h after the last inhibitor or placebo intake

SUMMARY:
This clinical phase I trial had 3 arms: inhibition by fluconazole, inhibition by ciprofloxacin and placebo. Subjects were treated for 3 days prior to the study day. The intervention was a single dose of 1 gram metamizole. We took blood samples at set time points and analysed the concentration of the main metabolites of metamizole at each time point in plasma.

DETAILED DESCRIPTION:
While the clinical pharmacokinetics of metamizole have been described in detail before, the enzymes responsible for the metabolism have not been identified yet (except for the acetylation of 4-aminoantipyrine). Former investigations delivered mixed results and the question of the participation of the hepatic cytochrome p450 enzymes could not been answered.

Thus, a double-blind randomized cross over clinical phase I study with healthy, male, caucasian volunteers was conducted. After giving consent for participation and enrolment, the subjects were treated for 3 days with either one inhibitor (either ciprofloxacin, CYP1A2 inhibitor, or fluconazole, strong CYP2C9 and moderate CYP2C19 and CYP3A4 inhibitor) or placebo. The doses were 750 mg ciprofloxacin twice daily for 3 days and in the morning of the study day or 400 mg fluconazole loading dose with consecutive 200 mg fluconazole once daily. For the study day, the subject were invited to the study center and a venous access was placed on the non-dominant arm. The last dose of either inhibitor or placebo was taken 1h prior to a single dose of 1000 mg metamizole. Blood samples were drawn at t: 0h, 0.25h, 0.5h, 0.75h, 1h, 2h, 3h, 4h, 6h, 8h, 12h and 24h. The blood samples were centrifuged, the plasma was isolated and frozen at -20°C. All subjects received both inhibitors and placebo treatment, attending to a total of 3 study days. Furthermore, the genotype for CYP1A2, CYP2B6, CYP2C9, CYP2C19 and CYP2D6 was assessed.

Plasma samples will be analyzed and the concentrations of the main metabolites of metamizole and the inhibitors will be measured. Pharmacokinetic parameters such as maximal concentration, half life, time to reach maximal concentration and the area under the curve will be assessed and compared.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 18 and 28 kg/m2 (inclusive) and bodyweight at least 50 kg at screening
* Systolic blood pressure: 100-140 mmHg, diastolic blood pressure: 60-90 mmHg and heart rate: 45-90 bpm (inclusive), measured on the leading arm*, in the supine position at screening
* No clinically significant findings on the physical examination on the physical examination at screening
* Signed informed consent prior to any study-mandated procedure
* Haematology and clinical chemistry results not deviating from the normal range to clinically relevant extent at screening
* Ability to communicate well with the investigator to understand and comply with the requirements of the study

Exclusion Criteria:

* Smoking > 5 cigarettes per day
* History or clinical evidence of alcoholism or drug abuse within the 3- year period prior to screening
* Loss of ≥ 250 ml of blood within 3 months prior to screening
* Treatment with an investigational drug within 30 days prior to screening
* Previous treatment with any prescribed or over the counter medication (including herbal medicines such as St John's Wort) within 2 weeks prior to the intended start of the study
* Legal incapacity or limited legal capacity at screening
* Positive results from urine drug screen at screening
* History or clinical evidence of any disease
* Known hypersensitivity to Metamizole (Novalgin®), ciprofloxacin (Ciproxin®), fluconazole (Diflucan®) or any other excipients in the drug formulation

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Assessment of the area under the plasma concentration vs time (AUC) | Study day (24 hours)
  Assessment of the change in AUC of the main metabolites of metamizole (4-methylaminoantipyrine, 4-aminoantipyrine, 4-acetylaminoantipyrine and 4-formylaminoantipyrine) in the 3 arms
Assessment of peak plasma concentration (Cmax) | Study day (24 hours)
  Assessment of the change of Cmax of the main metabolites of metamizole (4-methylaminoantipyrine, 4-aminoantipyrine, 4-acetylaminoantipyrine and 4-formylaminoantipyrine) in the 3 arms
Assessment of the time to reach peak plasma concentration (tmax) | Study day (24 hours)
  Assessment of the change in tmax of the main metabolites of metamizole (4-methylaminoantipyrine, 4-aminoantipyrine, 4-acetylaminoantipyrine and 4-formylaminoantipyrine) in the 3 arms
Assessment of the half-life (t1/2) | Study day (24 hours)
  Assessment of the change in t1/2 of the main metabolites of metamizole (4-methylaminoantipyrine, 4-aminoantipyrine, 4-acetylaminoantipyrine and 4-formylaminoantipyrine) in the 3 arms

SECONDARY OUTCOMES:
Compliance to the Pretreatment with Ciprofloxacin and Fluconazole | Study day (24 hours)
  Assessment of the area under the plasma concentration vs time of ciprofloxacin and fluconazole on the study day

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bachmann F, Duthaler U, Rudin D, Krahenbuhl S, Haschke M. N-demethylation of N-methyl-4-aminoantipyrine, the main metabolite of metamizole. Eur J Pharm Sci. 2018 Jul 30;120:172-180. doi: 10.1016/j.ejps.2018.05.003. Epub 2018 May 8. PMID 29746911
- [Result] Levy M, Zylber-Katz E, Rosenkranz B. Clinical pharmacokinetics of dipyrone and its metabolites. Clin Pharmacokinet. 1995 Mar;28(3):216-34. doi: 10.2165/00003088-199528030-00004. PMID 7758252